CLINICAL TRIAL: NCT04802941
Title: Optimizing Neoadjuvant Systemic Treatment for Breast Cancer by Clinical Decision Support System
Brief Title: Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center of Personalized Medicine, Pirogova (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other); I.M. Sechenov First Moscow State Medical University (Other); Novosibirsk Oncology Center (Unknown)
Responsible Party: Principal Investigator, Evgeny Pokushalov, Director for research and development, Center of Personalized Medicine, Pirogova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210312/2
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Decision Support Systems, Clinical
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Chemotherapy by CDSS (Experimental)
  Interventions: Device: Neoadjuvant Chemotherapy by CDSS (MedicBK)
- Neoadjuvant Chemotherapy in General practice (Active Comparator)
  Interventions: Drug: General practice

INTERVENTIONS:
Device: Neoadjuvant Chemotherapy by CDSS (MedicBK) — CDSS (MedicBK) captures the patient-specific data required to determine appropriate care decisions from the EMR and then presents relevant data alongside treatment suggestions to clinicians. MedicBK uses algorithms for presenting treatment suggestions framed by guideline-based therapy and personalized personalized evidence-based therapy. MedicBK consists of three main blocks: database, network meta-analysis, and heterogeneity of treatment effects assessment.
  Arms: Neoadjuvant Chemotherapy by CDSS
Drug: General practice — General practice
  Arms: Neoadjuvant Chemotherapy in General practice

SUMMARY:
This study compares two approaches of upfront chemotherapy in breast cancer.

DETAILED DESCRIPTION:
A Decision Support System (DSS) is an information system that supports business, medical, educational or organisational decision-making activities. DSSs fuse human knowledge and technology to support and improve decision-making.

The area of precision oncology that supports the treatment of breast cancer has not only seen an increase in the availability of different treatment choices but also genomic tools to support the decision-making process. CDSSs have been available for use in clinical oncology practice for over a decade. However, there has been some criticism around the utility of CDSS in personalised medicine decision-making of breast cancer, with these systems often viewed as aids better suited to support the 'average' patient's requirements rather than personalised treatment for the individual patient.

The purpose of the current study is to evaluate an innovative CDSS (MedicBK) platform based on the comparison of multiple treatments simultaneously in making care decisions taking into account the individual characteristics of patients, i.e., based on personalized evidence-based medicine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed infiltrating breast cancer
* Stage II or stage III disease. Nodal status must be examined by ultrasound, fine needle aspiration, sentinel node biopsy, or FDG-PET scan.
* Age ≥18
* Eastern Cooperative Oncology Group performance status ≤1
* Adequate bone marrow function (ANC >1.5 x 109/l, platelets >100 x 109/l)
* Adequate hepatic function (ALAT, ASAT and bilirubin <2.5 times upper limit of normal)
* Adequate renal function (creatinine clearance >50 ml/min)
* LVEF ≥50% measured by echocardiography or MUGA
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Absence of any medical condition that would place the patient at unusual risk.
* Signed written informed consent

Exclusion Criteria:

* previous radiation therapy or chemotherapy
* other malignancy except carcinoma in situ, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiation therapy.
* current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection
* evidence of distant metastases. Evaluation of the presence of distant metastases may include chest X-ray, liver ultrasound, isotope bone-scan, CT-scan of chest and abdomen and/or FDG-PET scan, according to local procedures.
* evidence of bilateral infiltrating breast cancer. Evaluation of the presence of bilateral infiltrating breast cancer may include mammography, breast ultrasound and/or MRI breast.
* concurrent anti-cancer treatment or another investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pathological complete response | at week 30
  To compare the efficacy of Neoadjuvant Chemotherapy in general practice and by CDSS

SECONDARY OUTCOMES:
Number of patients with grade >2 adverse events as a measure of safety and tolerability | up to week 35
  to describe the safety of the various regimens toxicity is compared between the two arms
identify prognostic and predictive for pathological complete response | within one year after end of treatment
  To identify prognostic and predictive for pathological complete response after neoadjuvant treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Evgeny Pokushalov, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided